CLINICAL TRIAL: NCT05174884
Title: A Phase 1 Clinical Trial to Evaluate the Pharmacokinetics, Removability, Safety, and Tolerability of Casea S Contraceptive Implants
Brief Title: Casea S Contraceptive Implants (Casea S) Trial
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1630531
Record Dates: First submitted 2021-08-25; First posted 2022-01-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Contraception
Keywords: Long Acting Reversible Contraceptive
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Casea S pellet (Experimental): In Part 1 of this study, four women will each have a single Casea S pellet (22.2 mg ENG) inserted into the inner aspect of the non-dominant upper arm.
  Interventions: Drug: 22.2 mg Etonogestrel (ENG)
- Two Casea S pellets (Experimental): In Part 2 of this study, sixteen women will each have two Casea S pellets (44.4 mg ENG) inserted into the inner aspect of the non-dominant upper arm.
  Interventions: Drug: 44.4 mg Etonogestrel (ENG)

INTERVENTIONS:
Drug: 22.2 mg Etonogestrel (ENG) — Subdermal insertion of a single Casea S pellet (22.2 mg ENG) in healthy female participants
  Other Names: Casea S
  Arms: Single Casea S pellet
Drug: 44.4 mg Etonogestrel (ENG) — Subdermal insertion of a two Casea S pellet (44.4 mg ENG) in healthy female participants
  Other Names: Casea S
  Arms: Two Casea S pellets

SUMMARY:
This is a single-center, two-part, Phase 1 study to evaluate the pharmacokinetics (PK) of ENG, removability, safety, and tolerability of Casea S pellets inserted subdermally in healthy women of reproductive age. The goal is to select for further investigation a dose of Casea S that is both safe and has a PK profile consistent with contraceptive protection for at least 78 weeks.

DETAILED DESCRIPTION:
In Part 1 of this study, four women will each have a single Casea S pellet (22.2 mg ENG) inserted into the inner aspect of the non-dominant upper arm after a negative urine pregnancy test. The insertion site and pellet location will be verified, marked, and photographed. ISRs and AEs will be assessed.

In Part 2 of this study, approximately sixteen women will each have two Casea S pellets (44.4 mg ENG) inserted into the inner aspect of the non-dominant upper arm. The insertion site and pellet location will be verified, marked, and photographed. ISRs and AEs will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Participants may be included in the study if they meet all of the following criteria:

* willing and able to provide signed informed consent
* female between 18 to 45 years of age (inclusive)
* healthy based on results of medical evaluation including medical history, vital signs, and physical exam
* has regular menstrual cycle (21 to 35 days)
* not at risk for pregnancy (i.e., sterilized)
* has a Body Mass Index (BMI) of 18 to 29.9
* provides normal mammogram results within the last year before enrollment for women 40 or older
* is willing and able to comply with all study requirements and return to the investigational site for the follow-up procedures and assessments as specified in this protocol
* Part 2 participants only: has daily access to a smartphone, tablet, or computer with internet access.

Exclusion Criteria:

Participants will be excluded from participating in this study if they meet any of the following criteria:

* has multiple risk factors for cardiovascular disease (e.g., smoking, diabetes, obesity, hypertension, high LDL (low density lipoprotein), or high triglyceride levels)
* has current or history of ischemic heart disease or cerebrovascular disease
* has current or previous thromboembolic disorders
* has systemic lupus erythematosus
* has rheumatoid arthritis on immunosuppressive therapy
* has migraine with aura
* has undiagnosed abnormal vaginal bleeding
* has known or suspected breast cancer, history of breast cancer or other progestin-sensitive cancer
* has current or history of cervical cancer
* has cirrhosis, liver tumors (benign or malignant), or active liver disease
* has one or more baseline liver function test(s) above the local laboratory's normal range
* has a hemoglobin <10.5 g/dL
* has used any injectable contraceptive in the past 6 months
* has used any of the following medications within 4 weeks before enrollment:

  * any investigational drug
  * prohibited drugs (listed in Section 6.3.3.4.4.1 of the study protocol)
  * oral contraceptives, contraceptive ring, or patch
  * levonorgestrel intrauterine device (LNG IUD) or contraceptive implant
* is pregnant
* is currently breastfeeding
* desires to become pregnant in the subsequent 30 months
* has been pregnant in last 3 months
* is using or planning to use prohibited drugs for their intended study duration
* has abnormal cervical cytology requiring treatment
* has known sensitivity to ENG
* plans to move to another location in the next 30 months
* is participating in any other clinical trial with a biomedical intervention
* has any condition (social or medical), that in the opinion of the site investigator would make study participation unsafe, would interfere with adherence to the clinical study requirements, or complicate data interpretation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) | 12 weeks; 52 weeks; 114 weeks
  Maximum observed serum concentration (Cmax) measured by blood samples collected at multiple timepoints before and after pellet insertion
Time to Cmax (tmax) | 12 weeks; 52 weeks; 114 weeks
  Time to Cmax (tmax) measured by blood samples collected at multiple timepoints before and after pellet insertion
Geometric mean serum ENG concentration | 28 days; 114 weeks
  Geometric mean serum ENG concentration at treatment days 28 and 84
Area under concentration time curve (AUC 0-28) | 28 days; 154 days; 364 days
  Area under the concentration time curve through days 28 and day 84
Predicted concentration at day 546 and probability of exceeding 90 pg/mL through day 546 | 52 weeks
  pharmacokinetics of ENG after subdermal insertion of 2 Casea S pellets
Assessment of the removability of Casea S pellets | up to 52 weeks
  Number and descriptions of incidence of removal complications
Assessment Casea S pellets removability | up to 52 weeks
  Time of the procedure duration of procedure
Ability to completely remove the pellet and ease of removal | up to 52 weeks
  Physician's assessment of the removability of Casea S pellets qualified as "complete removal, partial removal, or not removed" on the study removal assessment.
Time to undetectable ENG levels | 114 weeks
  Apparent absorption half-life; Predicted concentration at day 546 and probability of exceeding 90 pg/mL through day 546; Time above 90 pg/mL

SECONDARY OUTCOMES:
Occurrence of treatment emergency adverse events, significant changes in vital signs, weight, vaginal bleeding patterns and perceptions, abnormalities in serum chemistry, occurrence of implant site reactions | up to 114 weeks
  Safety and tolerability of Casea S pellets measured by the occurrence of treatment emergency adverse events, significant changes in vital signs, weight, vaginal bleeding patterns and perceptions, abnormalities in serum chemistry, occurrence of implant site reactions
Assessment of the ease of insertion of Casea S pellets | up to 114 weeks
  Physician's report of success and ease of insertion. Ease of insertion qualified as "easy, moderate, or difficult" on the study insertion assessment.
Assessment of the duration of Casea S pellets insertion | up to 114 weeks
  Time of the procedure duration
Assessment of the complications of insertion of Casea S pellets | up to 114 weeks
  Number and descriptions of the incidence of insertion complications.
Follicular and luteal activity following subdermal insertion of Casea S pellets | up to 114 weeks
  Estradiol (E2) and progesterone (P4) levels
Estimate of ENG release rates using explant analysis | up to 114 weeks
  Cumulative amount of ENG released over time, average daily release in 3 months and up to 130 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Nanda, M.D., Principal Investigator — FHI 360
Locations (1):
- Clinica Profamilia, Santo Domingo, DN, Dominican Republic

IPD SHARING:
Plan to Share IPD: No